CLINICAL TRIAL: NCT05409690
Title: Value of Renal Resistive Arterial Index for Differential Diagnosis of Patient With Anticipated Acute Kidney Injury Administered to Emergency Department
Brief Title: Renal Arterial Resistive Index for Differential Diagnosis of Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Bedriye Muge Sonmez, asossicated professor, Ankara Diskapi Training and Research Hospital
Other Study IDs: AnkaraDiskapiTRHAKI
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; renal resistive index; doppler ultrasound
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
early differential diagnosis of anticipated acute kidney injury via ultrasound renal resistive index calculation

DETAILED DESCRIPTION:
acute kidney injury is a common clinical syndrome introducing to emergency services with varying symptoms. acute kidney injury is divided into 3 subgroups: prerenal, renal and postrenal. there is not any certain laboratory or imaging modality for early detection of injury's type. calculation of renal resistive index with doppler ultrasound at emergency setting can be helpful for early detection of etiology of acute kidney injury subgroup.patient will be selected according to clinical status and detailed history and laboratory parameters.renal resistive index will we calculated with doppler ultrasound of arcuate and interlober arteries of kidneys. resistive index values of acute kidney injury patients will be compared depending on further tests and resistive indexes of suggestive etiologies will be compared according to final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18
2. patient with acute kidney injury diagnosed according to KDIGO, AKIN or RIFLE criteria

Exclusion Criteria:

1. end stage kidney disease
2. patients receiving renal replacement treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient administering to emergency service with acute kidney injury independent of etiology
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-11-10 (Estimated)

PRIMARY OUTCOMES:
increased resistive index | time spent at emergency service until renal doppler is done and resisitive index is calculated (6 hours)
  differential diagnosis of acute kidney injury using renal doppler ultrasound and resistive index and comparison of subgroups

SECONDARY OUTCOMES:
mortality | mortality at 7 days
  mortality
mortality | mortality at 28 days
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Research and Training Hospital, Ankara, Turkey (Türkiye)